CLINICAL TRIAL: NCT01510639
Title: Results of Subacromial Surgery; The Influence of Growth Factors (PDGF), Applied as Autologous Thrombocyte Concentrate, on Functional Recovery
Brief Title: The Influence of Growth Factors (PDGF), Applied as Autologous Thrombocyte Concentrate, on Functional Recovery
Acronym: PRP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Dr. N. Wolterbeek, Study Coordinator, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-08.05A/PDGF; NL19106.100.07 (Other: CCMO)
Record Dates: First submitted 2012-01-09; First posted 2012-01-16 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Rotator Cuff Rupture; Subacromial Impingement
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cuff repair PRP (Experimental): Cuff repair Platelet Rich Plasma: The application of autologous thrombocyte concentrate in the cuff repair group
  Interventions: Biological: Platelet Rich Plasma
- Cuff repair Control (No Intervention): No intervention
- NEER PRP (Experimental): Neer Platelet Rich Plasma: The application of autologous thrombocyte concentrate in the NEER surgery group
  Interventions: Biological: Platelet Rich Plasma
- NEER Control (No Intervention): No intervention

INTERVENTIONS:
Biological: Platelet Rich Plasma — The application of autologous thrombocyte concentrate (PRP). This is a concentrate with a high amount of thrombocytes (containing growth factors), obtained by centrifuging the patient's own blood. The concentrate is applied into the subacromial space after closure.
  Arms: Cuff repair PRP; NEER PRP

SUMMARY:
The purpose of this study is to test the hypothesis that the application of PRP leads to faster wound healing, less wound healing disorders, less pain and faster functional recovery after subacromial surgery.

DETAILED DESCRIPTION:
Subacromial surgery of the shoulder is performed often. It concerns space creating interventions (open and arthroscopic subacromial decompression) and rotator cuff surgery (open and arthroscopic). In this kind of surgery good wound healing and tissue recovery is of great importance to achieve optimal results. Wound healing disorders, pain and the formation of adhesions may negatively influence the postoperative course and lead to extended rehabilitation. This has an unfavourable influence on the personal well being of the patient and the possibility to return to labour. Especially in cuff surgery the course is strongly influenced by the healing of the attachment of the cuff to the bone. Besides the development of minimal invasive techniques, it's necessary to look for possibilities to decrease the morbidity of these procedures. Recent studies show that growth factors play a major role in wound healing. This concerns particularly TFG-B (transforming growth factor B) and PDGF (platelet derived growth factor) present in thrombocytes. They act as chemotactic agents for polymorphonuclear leucocytes, macrophages, fibroblasts and lymphocytes. Both growth factors stimulate the wound healing and cause improved angiogenesis and fibroplasia. They also play a role in wound retraction and remodelling. In animal-experimental models it is proved that the application of TGF-B and PDGF improves woundhealing and leads to better mechanical properties of the scar tissue. Faster and better wound healing and decreased development of adhesions after subacromial surgery can possibly be influenced favourably by using thrombocyte concentrate. In the treatment with autologous thrombocyte concentrate a thrombocyte rich concentrate is obtained by a centrifuging method (Gravitational Platelet System (GPS), Biomet, Warsaw USA) (platelet rich plasma or PRP), that can be applied in the operating field. The concentrate is harvest from the patients own blood, sampled during the procedure. At random the concentrated is applicated and both groups are compared postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Given informed consent
* Clinical indication for Arthroscopic Sub-acromial decompression, i.e.: Painful arc, pain at abduction, positive Hawkinstest Insufficient clinical improvement after (at least) 6 months of conservative treatment or Clinical indication for a arthroscopic cuff repair of a MRI-proven treatable rotator cuff tear.

Exclusion Criteria:

* Coagulopathy
* Thrombocytopenia
* Use of corticosteroids
* Diabetics Mellitus
* Omarthritis
* AC-arthrosis
* Cuff arthropathy
* Neurological deficit at the ipsi-lateral extremity
* (Wish for) Pregnancy
* VAS <2 or VAS >9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-07; Primary Completion 2013-07 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in VAS pain | 2 years
  Change in painscore measured on a VAS scale

SECONDARY OUTCOMES:
Functional recovery | 2 years
  Several questionnaires (RAND-36, SST, and Constant score) and functional tests are measured (Range of motion)
The amount of patients that had adequate wound healing | 2 years
  At different follow-up moments would healing is evaluated (6 weeks - 12 weeks - 1 year - 2 years)
The amount of patient who were able to resume their work | 2 years
  At different follow-up moments it is evaluated if patients was able to resume work (6 weeks - 12 weeks - 1 year - 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Petra E Flikweert, drs, Principal Investigator — St Antoniusziekenhuis; Gie Auw yang, Dr, Principal Investigator — St. Antoniusziekenhuis; Jacco Zijl, drs, Principal Investigator — St. Antoniusziekenhuis
Locations (1):
- st. Antoniusziekenhuis, Nieuwegein, Netherlands